CLINICAL TRIAL: NCT00672542
Title: Phase I Study of Active Immunotherapy of Metastatic Melanoma With Mature Autologous Dendritic Cells Transfected With Tumor Antigen RNA and Small Inhibitory RNAs to Alter Proteasomal Antigen Processing
Brief Title: Immunotherapy of Melanoma With Tumor Antigen RNA and Small Inhibitory RNA Transfected Autologous Dendritic Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scott Pruitt (Other)
Responsible Party: Sponsor-Investigator, Scott Pruitt, Associate Professor of Surgery, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000806; IND # BB-13545; NIH OBA # 0708-874
Record Dates: First submitted 2008-02-03; First posted 2008-05-06 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Metastatic Melanoma; Absence of CNS Metastases
Keywords: melanoma; dendritic cell; immunoproteasome; vaccine
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Vaccination with melanoma tumor associated antigen RNA loaded dendritic cells derived from untreated monocytes
  Interventions: Biological: Proteasome siRNA and tumor antigen RNA-transfected dendritic cells
- B (Experimental): Vaccination with melanoma tumor associated antigen RNA loaded dendritic cells derived from monocytes transfected with control siRNA
  Interventions: Biological: Proteasome siRNA and tumor antigen RNA-transfected dendritic cells
- C (Experimental): Vaccination with melanoma tumor associated antigen RNA loaded dendritic cells derived from monocytes transfected with siRNA targeting the three inducible immunoproteasome subunits
  Interventions: Biological: Proteasome siRNA and tumor antigen RNA-transfected dendritic cells

INTERVENTIONS:
Biological: Proteasome siRNA and tumor antigen RNA-transfected dendritic cells — The safety and toxicity of vaccination with tumor antigen RNA-transfected dendritic cells (DC), derived from either untransfected or siRNA-transfected monocytes, will be evaluated in subjects with metastatic melanoma. Subjects will undergo leukapheresis and monocytes will be isolated. These monocytes will then be left untreated (Study Arm A) or transfected with either control siRNA (Study Arm B) or siRNA targeting immunoproteasome subunits LMP2, LMP7, and MECL1 (Study Arm C), then differentiated into DC in vitro . After the induction of maturation, these DC will be transfected with RNA encoding defined melanoma antigens MART, MAGE-3, tyrosinase, and gp100. These RNA-transfected autologous DC will be cryopreserved, then used to vaccinate subjects with metastatic melanoma, each of whom will receive a total of six intradermal (ID) injections using 1x10e7 DC at each cycle, administered weekly.

SUMMARY:
Transfection with siRNA targeting the immunoproteasome alters proteasome-mediated antigen processing by the dendritic cell, generating TAA-derived peptides that we hypothesize, based on preclinical results, will induce enhanced anti-melanoma immune responses. This phase I study, open to subjects with metastatic melanoma, will assess the safety of vaccination with melanoma tumor associated antigen-encoding RNA-transfected mature dendritic cells derived from monocytes that have been either untreated, transfected with control siRNA, or transfected with siRNA targeting the inducible immunoproteasome beta subunits LMP2, LMP7, and MECL1. A combination of RNAs encoding melanoma tumor associated antigens MART-1, tyrosinase, gp100, and MAGE-3 will be utilized for dendritic cell transfection. The vaccine will be administered by intradermal injection in the extremities. Clinical and laboratory toxicities will be characterized for each study arm. As a secondary objective, this phase I study will also assess the anti-melanoma immune responses, as well as clinical responses, induced by vaccination with this dendritic cell-based product.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed metastatic melanoma.
* Karnofsky performance status greater than or equal to 70%.
* Estimated life expectancy > 6 months.
* Age > 18 years.
* Adequate hematologic function
* Adequate renal and hepatic function
* Ability to understand and provide signed informed consent that fulfills Institutional Review Board guidelines.
* Ability to return to Duke University Medical Center for adequate follow-up as required by this protocol.

Exclusion Criteria:

* Subjects undergoing concurrent chemotherapy, radiation therapy, or immunotherapy will be excluded.
* The subject has previously irradiated, surgically treated, or newly diagnosed central nervous system (CNS) metastases will be excluded (Pre-enrollment head CT is not required if not indicated by clinical signs or symptoms).
* Subjects with a history of autoimmune disease such as, but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis will be excluded.
* Subjects with serious concurrent chronic or acute illness such as pulmonary (asthma or COPD), cardiac (NYHA class III or IV) or hepatic disease, or other illness considered by the principal investigator to constitute an unwarranted high risk for investigational drug administration will be excluded.
* Subjects with medical or psychological impediment to probable compliance with the protocol will be excluded.
* Subjects with concurrent second malignancy other than melanoma or non-melanoma skin cancer will be excluded. In the event of prior non-melanoma malignancies treated surgically, the subject must be considered NED (no evidence of disease) for a minimum of 3 years prior to enrollment.
* Presence of an active acute or chronic infection, including symptomatic urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot) or viral hepatitis (as determined by HBsAg and Hepatitis C serology) will lead to subject exclusion.
* Subjects receiving steroid therapy (or other immunosuppressive agents such as azathioprine or cyclosporine A) are excluded on the basis of potential immune suppression.
* Subjects with inadequate peripheral vein access to undergo leukapheresis will be excluded.
* Female subjects with a positive pregnancy test, as well as those who have not previously undergone hysterectomy and/or bilateral oophorectomy and are unwilling to utilize a medically approved form of contraception, from the time of enrollment until 6 weeks after the final immunization, will be excluded.
* Male subjects, not previously surgically sterilized, who are unwilling to use a condom with spermicide during any sexual activity occurring over the entire immunization period and for the 6 weeks that immediately follow the final immunization will be excluded.
* Subjects with a documented history of severe allergic reaction to beta-lactams, eggs or soy products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-01; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
For this Phase I study, subjects will be evaluated both clinically and with laboratory testing for any signs of toxicity associated with vaccination. | 3 months after last vaccination

SECONDARY OUTCOMES:
For each subject, the induction of anti-melanoma immune responses will be assessed by in vitro testing. | At least 3 months after final vaccination
For each subject, clinical responses to vaccination will also be assessed. | At least 3 months, and up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott K Pruitt, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Dannull J, Haley NR, Archer G, Nair S, Boczkowski D, Harper M, De Rosa N, Pickett N, Mosca PJ, Burchette J, Selim MA, Mitchell DA, Sampson J, Tyler DS, Pruitt SK. Melanoma immunotherapy using mature DCs expressing the constitutive proteasome. J Clin Invest. 2013 Jul;123(7):3135-45. doi: 10.1172/JCI67544. Epub 2013 Jun 24. PMID 23934126